CLINICAL TRIAL: NCT03020498
Title: Protective Mechanisms Against a Pandemic Respiratory Virus. Project 1: B-cell Immunity to Influenza. Technical Development Project 1: Measuring the Immunome: Genomic Approaches to B-cell Repertoire - Years 2 (2010) & 3 (2011)
Brief Title: B-cell Immunity to Influenza (SLVP017) - Years 2 (2010) & 3 (2011)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Study Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-17218-2010-2011; 2U19AI057229-06 (NIH)
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: Inactivated influenza vaccine; Live, attenuated influenza vaccine; Child identical twins and non-twins; Young and elderly non-twin adults
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A: 8-17 yo identical twins (Other): Group A: 8-17 year-old identical twin pairs randomly assigned to Fluzone (trivalent, inactivated influenza vaccine (TIV)) or FluMist (live, attenuated influenza vaccine (LAIV)) within the pair
  Interventions: Biological: Fluzone; Biological: FluMist
- Group B: 8-30 yo non-twin (Other): Group B: 8-30 years old non-twin individuals randomly assigned to Fluzone (trivalent, inactivated influenza vaccine (TIV)) or FluMist (live, attenuated influenza vaccine (LAIV))
  Interventions: Biological: Fluzone; Biological: FluMist
- Group C: 70-100 yo non-twin (Other): Group C: 70-100 years old non-twin elderly adults given Fluzone (trivalent, inactivated influenza vaccine (TIV))
  Interventions: Biological: Fluzone

INTERVENTIONS:
Biological: Fluzone — Influenza Virus Vaccine Suspension for Intramuscular Injection
Biological: FluMist — Influenza Virus Vaccine Live, Intranasal Intranasal Spray
  Arms: Group A: 8-17 yo identical twins; Group B: 8-30 yo non-twin

SUMMARY:
In this exploratory study, investigators will be looking at immune response differences between age groups and between the two different influenza vaccines given to identical twins, vaccine-naive young adults and elderly participants.

DETAILED DESCRIPTION:
This is an exploratory study of healthy children and adults who are given either standard trivalent, inactivated influenza vaccine (TIV) or live, attenuated influenza vaccine (LAIV). There are no exclusions for gender, ethnicity or race. Following confirmation of written informed consent, baseline blood samples will be drawn from all study participants prior to immunization. The volunteers enrolled in any the three groups (A,B,C) cannot have been immunized with previous year's seasonal influenza vaccine. The identical twins in Groups A will be randomized to each receive a different vaccine (TIV or LAIV) than their twin. The non-twin children in Group B will also be randomly assigned to receive either TIV or LAIV. Non-twin elderly adults in Group C will be given standard TIV. All participants will receive a single dose of their assigned influenza vaccine, either by intramuscular (IM) injection (TIV) or intranasal application (LAIV).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, ambulatory 8-17 year old identical twins, 8-30 year old non-twins, or 70-100 year old elderly non-twin adults.
2. Willing to complete the informed consent process.
3. Availability for follow-up for the planned duration of the study at least 28 days after immunization.
4. Acceptable medical history by medical history and vital signs.

Exclusion Criteria:

1. Prior vaccination with seasonal TIV or LAIV or H1N1.
2. Prior off-study vaccination with the current seasonal TIV or LAIV
3. Allergy to egg or egg products, or to vaccine components
4. Life-threatening reactions to previous influenza vaccinations
5. Asthma or history of wheezing
6. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
7. History of immunodeficiency (including HIV infection)
8. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
9. Blood pressure >150 systolic or >95 diastolic at first study visit
10. Hospitalization in the past year for congestive heart failure or emphysema.
11. Chronic Hepatitis B or C.
12. Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible in all groups; inhaled steroid use is not permissible except for non-LAIV Group C only). Use of oral steroids (<20mg prednisone-equivalent/day) may be acceptable for volunteers 70-100 yrs of age after review by the investigator.
13. Participants in close contact with anyone who has a severely weakened immune system should not receive LAIV (Groups A and B only)
14. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
15. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
16. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
17. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg. per day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
18. Receipt of blood or blood products within the past 6 months
19. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
20. Inactivated vaccine 14 days prior to vaccination
21. Live, attenuated vaccine within 60 days of vaccination
22. History of Guillain-Barré Syndrome
23. Pregnant or lactating woman
24. Use of investigational agents within 30 days prior to enrollment
25. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment
26. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Harry Greenberg, MD, Principal Investigator — Stanford University; Stephen Quake, PhD, Principal Investigator — Stanford University; Xiaosong He, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sasaki S, Holmes TH, Albrecht RA, Garcia-Sastre A, Dekker CL, He XS, Greenberg HB. Distinct cross-reactive B-cell responses to live attenuated and inactivated influenza vaccines. J Infect Dis. 2014 Sep 15;210(6):865-74. doi: 10.1093/infdis/jiu190. Epub 2014 Mar 27. PMID 24676204
- [Background] He XS, Holmes TH, Sanyal M, Albrecht RA, Garcia-Sastre A, Dekker CL, Davis MM, Greenberg HB. Distinct patterns of B-cell activation and priming by natural influenza virus infection versus inactivated influenza vaccination. J Infect Dis. 2015 Apr 1;211(7):1051-9. doi: 10.1093/infdis/jiu580. Epub 2014 Oct 21. PMID 25336731
- [Background] Brodin P, Jojic V, Gao T, Bhattacharya S, Angel CJ, Furman D, Shen-Orr S, Dekker CL, Swan GE, Butte AJ, Maecker HT, Davis MM. Variation in the human immune system is largely driven by non-heritable influences. Cell. 2015 Jan 15;160(1-2):37-47. doi: 10.1016/j.cell.2014.12.020. PMID 25594173
- [Derived] de Bourcy CFA, Dekker CL, Davis MM, Nicolls MR, Quake SR. Dynamics of the human antibody repertoire after B cell depletion in systemic sclerosis. Sci Immunol. 2017 Sep 29;2(15):eaan8289. doi: 10.1126/sciimmunol.aan8289. PMID 28963118

RESULTS

PARTICIPANT FLOW:
Groups:
- Group B: 8-30 yo Non-twin: Group B: 8-30 years old non-twin individuals given Fluzone (trivalent, inactivated influenza vaccine (TIV)) or FluMist (live, attenuated influenza vaccine (LAIV))
  Fluzone: Influenza Virus Vaccine Suspension for Intramuscular Injection
  FluMist: Influenza Virus Vaccine Live, Intranasal Intranasal Spray
Period: Overall Study
Arm/Group | Group A: 8-17 yo Identical Twins | Group B: 8-30 yo Non-twin | Group C: 70-100 yo Non-twin
Started | 14 | 41 | 36
Completed | 14 | 38 | 36
Not Completed | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: 8-17 yo Identical Twins | Group B: 8-30 yo Non-twin | Group C: 70-100 yo Non-twin | Total
Number analyzed (Participants) | 14 | 41 | 36 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.84 (3.53) | 21.82 (5.32) | 77.00 (5.313) | 42.27 (28.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 23 | 21 | 54
  Male | 4 | 18 | 15 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 0 | 7
  Not Hispanic or Latino | 12 | 36 | 36 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 13 | 0 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 12 | 22 | 36 | 70
  More than one race | 2 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 41 | 36 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Influenza Vaccine
Time Frame: Day 0 to 28
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 8-17 yo Identical Twins | Group B: 8-30 yo Non-twin | Group C: 70-100 yo Non-twin
Number analyzed (Participants) | 14 | 41 | 36
Participants | 14 | 38 | 36

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to 28 post-immunization
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 8-17 yo Identical Twins | Group B: 8-30 yo Non-twin | Group C: 70-100 yo Non-twin
Number analyzed (Participants) | 14 | 38 | 36
Participants | 1 | 1 | 1

3. Other Pre Specified Outcome: Investigate the Effects of Different Influenza Vaccines, Including Live Attenuated Vaccine (LAIV) and Inactivated Vaccine Delivered by Different Routes (Intranasal and IM), on B-cell Responses.
Time Frame: Day 0 to 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 0 to Day 28 of study participation
Description: Clinical Assessment performed at each visit
Arm/Group | Group A: 8-17 yo Identical Twins | Group B: 8-30 yo Non-twin | Group C: 70-100 yo Non-twin
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/38 | 0/36
Other Adverse Events (participants affected / at risk) | 1/14 | 1/38 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: 8-17 yo Identical Twins (N=14) | Group B: 8-30 yo Non-twin (N=38) | Group C: 70-100 yo Non-twin (N=36)
Light headedness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) — Reported after the blood draw.
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Reported during blood draw

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No